CLINICAL TRIAL: NCT01727583
Title: Boosting the Secretion of GLP-2 and GLP-1 Intestinal Hormones by Nutrients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 12.10.MET
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lipid 1 (Active Comparator): Meal intake
  Interventions: Dietary Supplement: meal intake
- Lipid-free (Placebo Comparator): Maltodextrine + proteins
  Interventions: Dietary Supplement: Placebo
- Lipid 2 (Active Comparator): Meal intake
  Interventions: Dietary Supplement: meal intake
- Lipid 3 (Active Comparator): Meal intake
  Interventions: Dietary Supplement: meal intake
- Lipid 4 (Active Comparator): meal intake
  Interventions: Dietary Supplement: meal intake

INTERVENTIONS:
Dietary Supplement: meal intake — Intake of meals characterized by lipid composition
  Arms: Lipid 1; Lipid 2; Lipid 3; Lipid 4
Dietary Supplement: Placebo
  Arms: Lipid-free

SUMMARY:
This pilot study is aimed at assessing the acute effect of several combinations of lipids differing in their fatty acid composition on glucagon-like-peptide (GLP)-2 and GLP-1 secretion in healthy subjects.

DETAILED DESCRIPTION:
In this study, the investigators aim to investigate the effect of various lipid types on GLP-2 and GLP-1 secretion. This will allow to determine the importance of lipids in nutritional solutions. Moreover, this will allow us to assess whether existing clinical formulas can be improved in order to stimulate GLP-2 and accelerate intestinal recovery.

ELIGIBILITY:
Inclusion Criteria:

* BMI : 19 - 24.9 kg.m-2
* Normal fasting glycemia
* Having obtained his informed consent.

Exclusion Criteria:

* Gastro-intestinal disease (ulcer), pancreatic disease, hepatic disease, metabolic diseases / disorders (diabetes, dyslipidemia), renal disease, cardiovascular disease (arterial hypertension), as determined by the medical screening visit and a blood analysis.
* Have had a gastrointestinal surgery (with the exception of appendices resection).
* Malabsorption disorders
* Lactose intolerance
* Significant weight loss during the past three months (more than 5% of initial weight)
* Have a regular consumption of medication
* Regular supplements (vitamins and minerals) intake during the previous month
* Have an alcohol intake: > 2 units a day
* Smoker (more than 2 cigarettes a day)
* Illicit substances intake, as stated on the medical screening questionnaire
* Allergy to any food or medication
* Anaemia defined by a number of erythrocytes or hemoglobin Hb or hematocrit Ht which are inferior to laboratory normal ranges
* Having given blood in the past three months or willing to give blood in the 3 months following the completion of the study
* Intense physical activity > 3 hours per week
* Currently participating or having participated in another clinical trial during the past month.
* Volunteer who cannot be expected to comply with the protocol, including consuming rapidly the study products, chronic medication intake

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
GLP-2 and GLP-1 kinetics | changes from baseline to 4 hours following meal intake
  GLP-2 and GLP-1 are measured using Elisa

SECONDARY OUTCOMES:
Intestinal and metabolic hormones | Changes from baseline to 4 hours following meal intake
  Those hormones will be measured based on enzymatic technics

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Principal Investigator — Nestlé / CDU / Metabolic Unit
Locations (1):
- Nestlé CDU / Metabolic Unit, Lausanne, Switzerland